CLINICAL TRIAL: NCT06690684
Title: Identification and Functional Study of Novel Biomarkers for Cardiovascular Diseases
Status: Enrolling by invitation | Type: Observational
Sponsor: Ya-Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Ya-Wei Xu, Shanghai 10th People's Hospital (Responsible Party), Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: Novel biomarkers 23K98
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Angiocardiography; Heart Failure; Ischemic Heart Disease; Acute Myocardial Infarction (AMI)
Keywords: angiocardiography; heart failure; ischemic heart disease; biomarkers; identification; function; Acute Myocardial Infarction (AMI)
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — BLOOD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PCI in patients with acute myocardial infarction
  Interventions: Biological: Hematological indicators; Biological: Serological indicators in patients with myocardial infarction; Biological: Levels of biomarkers in blood of patients with acute myocardial infarction

INTERVENTIONS:
Biological: Hematological indicators — This project is a retrospective clinical cohort study. STEMI patients undergoing PCI were selected to explore whether hematological indicators such as PIV, SHR, and Lp(a) can improve the accuracy of predicting short-term MACE events in STEMI patients.
Biological: Serological indicators in patients with myocardial infarction — This study selected STEMI patients who underwent PCI and collected their hematological indicators to explore the value of PIV, SHR, Lp(a) and other indicators in improving the accuracy of predicting MACE in STEMI patients in the short term.
Biological: Levels of biomarkers in blood of patients with acute myocardial infarction — Hemoglobin, neutrophil count, lymphocyte count, monocyte count and platelet count values, N-terminal pro-B type natriuretic peptide (NT-proBNP), peak creatine kinase isoenzymes (CK-MB), peak troponin T levels, total cholesterol (TC), fasting blood glucose (FBG), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C) and blood urine nitrogen, blood creatinine (Cr) and other indicators

SUMMARY:
Cardiovascular diseases, mainly represented by ischemic heart disease and heart failure, are the number one killers of human health today. The China Cardiovascular Health and Disease Report 2022 pointed out that the current number of people suffering from cardiovascular diseases in China is 330 million, and cardiovascular diseases account for the highest proportion of disease deaths among urban and rural residents. With the increase of the population and the progress of aging in recent years, the number of patients with cardiovascular diseases is still increasing. Level three prevention is an important part of the long-term management of patients with cardiovascular diseases. Early identification of high-risk groups among patients with cardiovascular diseases and individualized and accurate treatment can greatly reduce the probability of cardiovascular events in patients, improve the quality of life and prognosis of patients, and reduce overall medical economic expenditure. However, at present, there is still a lack of effective biological markers in clinical practice that can give patients accurate positioning in all aspects. In this project, we intend to carry out the following research: (1) Based on real-world cohort research and observation, through proteomics, genomics, transcriptomics, metabolomics, etc., we will explore biomarkers that can be used for the evaluation of cardiovascular diseases from peripheral serum samples of patients with cardiovascular disease (2) Based on true The cohort research observation in the real world clarifies the effectiveness of the biomarkers screened in the first part of the research content and the correlation with the prognosis of the disease (3) Through bioinformatics analysis and basic function research, the function of the selected biomarkers and the mechanism of action in the organism are clarified. This project is expected to provide new criteria and theoretical basis for the prognostic management of clinical cardiovascular diseases.

DETAILED DESCRIPTION:
In this project, we will plan to carry out the following research: (1) Based on real-world cohort study observations, explore biomarkers that can be used for tertiary prevention assessment of cardiovascular disease from peripheral serum samples of cardiovascular disease patients through proteomics, genomics, transcriptomics, metabolomics, etc.(2) Based on real-world cohort study observations, clarify the effectiveness of the biomarkers screened in the first part of the research content and their correlation with disease prognosis (3) Through bioinformatics analysis and basic functional research, Clarify the functions of the screened biomarkers and their mechanisms of action in vivo. This project is expected to provide new evaluation criteria and theoretical basis for clinical cardiovascular disease prognostic management.

The specific research plan is as follows:

1. Study population: Patients diagnosed with myocardial infarction or heart failure (NYHA II-IV)
2. Inclusion criteria: 1. Subjects must be 30 years old or older when signing the informed consent form. Subject type and disease characteristics: a. Patients diagnosed with myocardial infarction, Killip I-V, mainly due to myocardial infarction, emergency department or hospitalization b. (1). Patients diagnosed with heart failure, NYHAII-IV, who came to outpatient clinics or hospitalizations mainly due to heart failure (2). Received diuretics within 30 days before enrollment (3). Structural cardiac abnormalities based on any local imaging measurements within the past 12 months (latest screening), defined as at least one of the following: oLAD≥ 3.8 cm, LAA≥20 cm2, LAVI>30mL/m2, LVMI≥115g/m2 (MIN)/95g/m2 (MIN), septum thickness or posterior wall thickness ≥ 1.1 cm (4). Subjects in sinus rhythm: NT-proBNP≥300pg/mL (BNP≥100pg/mL) or subjects with atrial fibrillation (or if atrial fibrillation status is unknown): NT-proBNP≥900pg/mL (BNP≥300pg/mL).
3. Exclusion criteria: 1. eGFR<25mL/min/1.73m2 at the screening visit;2. Serum/plasma potassium>5.0mmol/L at the screening visit;3. Acute inflammatory heart disease occurred within 60 days before enrollment;4. Coronary artery bypass surgery occurred 90 days before enrollment;6. Stroke or transient ischemic attack occurred within 30 days before enrollment; 7. The investigator believes that the subject's symptoms may be caused by other reasons, such as the patient's symptoms of difficulty breathing may be caused by severe lung disease, anemia or obesity. Specifically, patients with only symptoms and no organic cardiac changes due to the following conditions were excluded;8 2 consecutive measurements taken at least 2 minutes apart at screening, systolic blood pressure (SBP) ≥160mmHg and not receiving ≥3 antihypertensive drugs or ≥180mmHg (regardless of treatment);9. Life-threatening or uncontrollable arrhythmia at screening, including but not limited to: sustained ventricular tachycardia, or atrial flutter with resting ventricular rate>110bpm;10. Symptomatic hypotension at screening (Mean systolic blood pressure <90mmHg) 11. Had a left ventricular assist device at screening;12. Had a history of hyperkalemia or acute renal failure for>7 consecutive days during MRA treatment;13. Pregnant or nursing (lactation) women, where pregnancy is defined as the woman's condition after conception until termination of pregnancy, and a confirmed positive urine or serum test result for human chorionic gonadotropin;14. Have liver dysfunction classified as Child-PughC at screening.
4. Study process: Enrolled patients will be divided into two groups: myocardial infarction group and heart failure group based on the enrolled disease. Patients in the two groups have received standardized reperfusion therapy + ischemic cardiomyopathy treatment and anti-heart failure treatment respectively since the start of the study. Patients will be collected once before the start of treatment. Each patient needs to complete an enrollment assessment at the time of enrollment, and follow-up needs to be completed every year during the treatment period until the endpoint event occurs, or 5-year follow-up is completed.
5. Clinical data collection content:

All patients were required to complete general conditions, laboratory tests and auxiliary tests at enrollment, and major cardiovascular events and readmission events related to cardiovascular diseases were recorded during the follow-up period.

General conditions include: height, weight, age, gender, BMI, blood pressure, heart rate Laboratory tests and auxiliary tests include: NT-proBNP, BNP, blood routine (white blood cell count (WBC), red blood cell count (RBC), hemoglobin (Hb), hematocrit, platelets, mean corpuscular hemoglobin content (MCH), mean corpuscular hemoglobin concentration (MCHC), mean corpuscular volume (MCV), corpuscular volume distribution width (RDW)), liver and kidney function (Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP), creatine kinase (CK), serum creatinine, eGFR, blood urea nitrogen, bilirubin, electrolytes (sodium, serum potassium), thyroid function, urine routine examination, glycosylated hemoglobin, cardiac color Doppler examination Biological sample testing includes: proteomics, genomics, transcriptomics, metabolomics, etc.

Major cardiovascular events: acute myocardial infarction, stroke, cardiovascular death

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 30 years old and older at the time of signing the informed consent form.

Subject type and disease characteristics:

1. Patients diagnosed with myocardial infarction, Killip I-V, mainly due to myocardial infarction, emergency department or hospitalization
2. (1). Patients diagnosed with heart failure, NYHAII-IV, who came to outpatient clinics or hospitalizations mainly due to heart failure (2). Received diuretics within 30 days before enrollment (3). Structural cardiac abnormalities based on any local imaging measurements within the past 12 months (latest screening), defined as at least one of the following: oLAD≥ 3.8 cm, LAA≥20 cm2, LAVI>30mL/m2, LVMI≥115g/m2 (MIN)/95g/m2 (MIN), septum thickness or posterior wall thickness ≥ 1.1 cm (4). Subjects in sinus rhythm: NT-proBNP≥300pg/mL (BNP≥100pg/mL) or subjects with atrial fibrillation (or if atrial fibrillation status is unknown): NT-proBNP≥900pg/mL (BNP≥300pg/mL).

Exclusion Criteria:

1. eGFR < 25 mL/min/1.73 m2 at the screening visit;
2. Serum/plasma potassium > 5.0 mmol/L at the screening visit;
3. Acute inflammatory heart disease within 60 days before enrollment;
4. Coronary artery bypass grafting within 90 days before enrollment;
5. Stroke or transient ischemic attack within 30 days before enrollment;
6. The researcher believes that the subject's symptoms may be caused by other reasons, such as the patient's dyspnea symptoms may be caused by severe lung disease, anemia or obesity. Specifically, patients with only symptoms and no organic cardiac changes were excluded due to the following circumstances: 7. Systolic blood pressure (SBP) ≥160 mmHg and not receiving ≥3 antihypertensive drugs or ≥180 mmHg (regardless of the treatment received) for 2 consecutive measurements at least 2 minutes apart at screening;

8. Life-threatening or uncontrollable arrhythmias at screening, including but not limited to: sustained ventricular tachycardia, or atrial flutter with a resting ventricular rate >110 bpm; 9. Symptomatic hypotension (average systolic blood pressure <90 mmHg ) during the screening period; 10. Left ventricular assist device installed at screening; 11. History of hyperkalemia or acute renal failure for more than 7 consecutive days during MRA treatment; 12. Pregnant or lactating (lactating) women, where pregnancy is defined as the state of a woman from conception until termination of pregnancy, and confirmed by a positive human chorionic gonadotropin urine or serum test result; 13. Liver dysfunction classified as Hild-Pugh grade C at screening.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction or heart failure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
MACE | From the time of hospital discharge until the event of specific outcome, death, or loss to follow up, maximum 5 years.
  The composite events include a composite of all-cause mortality (death due to any cause), cardiovascular mortality (death due to cardiac cause), and heart failure rehospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Jing 'an District, Shanghai City, Shanghai, Jing 'an District, China

IPD SHARING:
Plan to Share IPD: Undecided